CLINICAL TRIAL: NCT04282083
Title: ITANET -Registry: Multicentric Collection of Cases on Neuroendocrin Gastro-Entero-Pancreatic Tumors (Title in Local Language: ITANET -Registry: Raccolta Multicentrica Dei Casi di Tumore Neuroendocrino Gastro-Entero-Pancreatico)
Brief Title: Protocol ITANET - Registry
Status: Recruiting | Type: Observational
Sponsor: Italian Association Neuroendocrine Tumors (Network)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2020-02-03; First posted 2020-02-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Gastro-entero Pancreatic Neuroendocrine Tumors
Keywords: GEP-NETs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study with the aim to create an Italian database for the collection of data on diagnostic approach, therapy and follow up of patients affected by GEP-NET (gastro-enteric-pancreatic neuroendocrine tumours). Data for approximately 200 italian patients were already previously collected in the ENETS database (international database). ENETS decided to interrupt the collection of the data for an indefinite period. For this reason, through an amendment (number 1) to the protocol, ITANET (Italian Association Neuro-endocrine Tumors) decided to transfer the italian data into a national database and to go on with the collection/update of the data, in order not to lose important clinical information.

DETAILED DESCRIPTION:
Each participating site will have access through the reserved area of webpage https://itanetdb.fullcro.org/, for the data recording in a database which ITANET set-up for the participating sites in Italy.

The eligible patients, visited at each participating site, will be asked to adhere to the ITANET-project through a proper Informed Consent obtainment procedure.

Adequate procedures are described in the protocol amendment 1 (and in a proper Standard Operating Procedure) also for the management of the already collected data in the previous ENETS registry whose transferral/update/deletion in the ITANET database are well defined and regulated in order to respect and preserve the patients' rights.

The data will be collected in an pseudo-anonymised way. Each patient will be identified by a code.

The data management and quality check of the Italian data is deputed to ITANET. The data will be collected in a prospective way, both for the new diagnoses (first visits) and for the follow up visits of patients with already acquired diagnosis. For the patients with already acquired diagnosis, these diagnostic data can be collected retrospectively, but not earlier than 1 year from the date of informed consent signature.The enrolment will take place during the outpatient visit or at the time of the hospitalisation for the NET-related surgery.

Of course, considering the observational nature of the study, the follow up visits will be planned on the basis of each patient's clinical need, which is different patient by patient, according to the disease staging, the primary tumour location, the eventual surgery.

The data flow will be the following:

* The participating site records the data in the database, waiting to be validated;
* ITANET has the role to check the recorded data for completeness and coherence in order to decide whether:

  1. The data are acceptable: in this case the data will be validated;
  2. There are discrepancies: in this case a query will be sent to the related site in order to check, correct/explain where applicable and to resubmit the data. The process starts again until final validation.

The data will be collected yearly to provide several information, such as:

* Type of NETs followed by the reference national sites for the management of the study pathology;
* Tools used for the diagnosis definition and the disease staging;
* Therapeutic approach (surgical or medical);
* Disease trend during follow up.

ELIGIBILITY:
Inclusion Criteria:

* age> or = 18 years;
* histologically/cytologically proved diagnosis of NET OR diagnosis supported by a PET Gallium 68 positivity and by at least a contrastografic imaging of second level (CT scan or NMR);
* Diagnosis of GEP-NET not antecedent 1 year since the Informed Consent signature;
* Grading G1, G2, G3 according to the classification WHO 2019;
* Tumor origin in digestive apparatus (GEP NETs) or tumor of unknown origin;
* Signed Informed consent.

Exclusion Criteria:

* Known tumor origin different from digestive apparatus (GEP NETs);
* no evidence of histologically/cytologically proved diagnosis of NET OR diagnosis supported by a PET Gallium 68 positivity and by at least a contrastografic imaging of second level (CT scan or NMR);
* Diagnosis of GEP-NET antecedent 1 year since the Informed Consent signature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by gastro-entero pancreatic neuroendocrine or unknown primary tumor
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2019-05-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of GEP-NET in Italy | 3 years
Different localisations of primary GEP-NET | 3 years
Time between symptoms appearance and diagnosis of GEP-NET | 3 years
Type of used and available treatments (medical and surgical) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MASSIMO FALCONI, Principal Investigator — San Raffaele Hospital
Locations (37):
- Italy (37):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Clinica Pederzoli, Peschiera del Garda, Verona
  - AO Ospedali Riuniti, Ancona
  - Azienda Ospedaliera Universitaria Consorziale Policlinico, Bari
  - Azienda Ospedaliera Universitaria Policlinico S. Orsola Malpighi, Bologna
  - IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna
  - Ospedale Regionale di Bolzano, Bolzano
  - ASST Spedali Civili, Brescia
  - Presidio Ospedaliero A. Perrino, Brindisi
  - Istituto Oncologico del Mediterraneo, Catania
  - Azienda Ospedaliera Universitaria, Ferrara
  - Ospedale Policlinico S. Martino, Genova
  - Ospedale Santa Maria Goretti, Latina
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - San Raffaele Hospital, Milan
  - IRCCS Istituto Nazionale Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - AOU Policlinico-Modena, Modena
  - Ospedale San Gerardo, Monza
  - AO Cardarelli, Naples
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Policlinico Università Federico II, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Centro di Riferimento Regionale per i Tumori Rari dell'adulto Università degli Studi di Palermo, Palermo
  - Ospedale Santa Chiara, Pisa
  - AOUSL-IRCCS-Reggio Emilia, Reggio Emilia
  - Presidio Ospedaliero di Rho, Rho
  - Istituti Fisioterapici Ospitalieri, Roma
  - Ospedale San Filippo Neri, Roma
  - Policlinico Umberto I, Roma
  - Sant'Andrea Hospital, Rome
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Universitaria, Sassari
  - Center for Immuno-Oncology Medical Oncology and Immunotherapy University of Siena, Siena
  - Azienda Ospedaliero Universitaria Città della salute e della Scienza, Torino
  - Ospedale Santa Chiara, Trento
  - Azienda Ospedaliera Universitaria integrata, Verona

REFERENCES:
- [Derived] Panzuto F, Partelli S, Campana D, de Braud F, Spada F, Cives M, Tafuto S, Bertuzzi A, Gelsomino F, Bergamo F, Marcucci S, Mastrangelo L, Massironi S, Appetecchia M, Filice A, Badalamenti G, Bartolomei M, Amoroso V, Landoni L, Rodriquenz MG, Valente M, Colao A, Isidori A, Fanciulli G, Bollina R, Ciola M, Butturini G, Marconcini R, Arvat E, Cinieri S, Berardi R, Baldari S, Riccardi F, Spoto C, Giuffrida D, Gattuso D, Ferone D, Rinzivillo M, Bertani E, Versari A, Zerbi A, Lamberti G, Lauricella E, Pusceddu S, Fazio N, Dell'Unto E, Marini M, Falconi M. Epidemiology of gastroenteropancreatic neuroendocrine neoplasms: a review and protocol presentation for bridging tumor registry data with the Italian association for neuroendocrine tumors (Itanet) national database. Endocrine. 2024 Apr;84(1):42-47. doi: 10.1007/s12020-023-03649-4. Epub 2024 Jan 4. PMID 38175391